CLINICAL TRIAL: NCT01909752
Title: Randomized Phase II Trial of Cyclophosphamide With Allogeneic Non-Small Cell Lung Cancer (NSCLC) DRibble Vaccine Alone or With Granulocyte-Macrophage Colony-Stimulating Factor or Imiquimod for Adjuvant Treatment of Definitively-Treated Stage IIIA or IIIB NSCLC
Brief Title: Combination Vaccine Immunotherapy (DRibbles) for Patients With Definitively-Treated Stage III Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UbiVac (Industry)
Collaborators: National Cancer Institute (NCI) (NIH); Providence Cancer Center, Earle A. Chiles Research Institute (Other); Providence Health & Services (Other); Mayo Clinic (Other); Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UbiVac DPV-001; R44CA121612 (NIH)
Record Dates: First submitted 2013-07-24; First posted 2013-07-26 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Lung cancer; DRibble Vaccine; Imiquimod; GM-CSF; HPV vaccine (Ceravix); Cyclophosphamide
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Cyclophosphamide; Imiquimod; Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim; Papillomavirus Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- DRibble Vaccine Alone (Experimental): Cyclophosphamide (300 mg/m2) will be administered as a single dose three days prior to beginning vaccine therapy. DRibble vaccine will be administered at Weeks 1, 4, 7, 10, 13, 16, 19, 25, 31, 37, and 43. Immunization with HPV vaccine intramuscular injection at the time of the first and third vaccinations.
  Interventions: Drug: Cyclophosphamide; Biological: DRibble vaccine; Biological: HPV vaccine
- DRibble vaccine with imiquimod (Experimental): Cyclophosphamide (300 mg/m2) will be administered as a single dose three days prior to beginning vaccine therapy. DRibble vaccine will be administered at Weeks 1, 4, 7, 10, 13, 16, 19, 25, 31, 37, and 43. Imiquimod cream (5%, 250 mg containing 12.5 mg imiquimod - one packet/day) will be self applied once per day starting with the second vaccine (week 4) and for four days following each vaccine cycle. Immunization with HPV vaccine intramuscular injection at the time of the first and third vaccinations.
  Interventions: Drug: Cyclophosphamide; Biological: DRibble vaccine; Drug: Imiquimod; Biological: HPV vaccine
- DRibble vaccine with GM-CSF (Experimental): Cyclophosphamide (300 mg/m2) will be administered as a single dose three days prior to beginning vaccine therapy. DRibble vaccine will be administered at Weeks 1, 4, 7, 10, 13, 16, 19, 25, 31, 37, and 43. GM-CSF will be administered at 50 mcg/day starting with the second vaccine (week 4) and continuing with each subsequent vaccine. Immunization with HPV vaccine intramuscular injection at the time of the first and third vaccinations.
  Interventions: Drug: Cyclophosphamide; Biological: DRibble vaccine; Drug: GM-CSF; Biological: HPV vaccine

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide (300 mg/m2) will be administered as a single dose three days prior to beginning vaccine therapy.
  Other Names: Cytoxin
Biological: DRibble vaccine — DRibble vaccine will be administered at Weeks 1, 4, 7, 10, 13, 16, 19, 25, 31, 37, and 43.
Drug: Imiquimod — Imiquimod cream (5%, 250 mg containing 12.5 mg imiquimod - one packet/day) will be self applied once per day starting with the second vaccine (week 4). Immediately following vaccination and for four days following each vaccine cycle (total 5 days) imiquimod will be applied to a 4 x 5-cm outlined area of healthy extremity skin that includes the vaccine site.
  Other Names: Aldara
  Arms: DRibble vaccine with imiquimod
Drug: GM-CSF — GM-CSF will be administered at 50 mcg/day starting with the second vaccine (week 4) and continuing with each subsequent vaccine. A volume of 0.2 cc will be delivered by the CADD-MSTM 3 Ambulatory infusion pump at a rate of 0.008 cc/hr. The pump will be refilled after three days for a total of six days of infusion.
  Other Names: Leukine
  Arms: DRibble vaccine with GM-CSF
Biological: HPV vaccine — Immunization with HPV vaccine will consist of two 0.5-mL intramuscular injection at the time of the first and third vaccinations. The preferred site of administration is the deltoid region of the upper arm.
  Other Names: Ceravix

SUMMARY:
This study will test an investigational vaccine, called DRibbles, for the treatment of non-small cell lung cancer (NSCLC). We hypothesize that vaccination with the DRibble vaccine will cause an immune responses against proteins contained in the DRibble vaccine and the protein antigens targeted by this strong immune response will include common antigens shared by both the vaccine and the patient's tumor.

DETAILED DESCRIPTION:
This is an open-label, randomized study in which the first 33 patients will be assigned to receive the either:

* DRibbles vaccine and HPV vaccine
* DRibbles vaccine, HPV vaccine, and imiquimod
* DRibbles vaccine, HPV vaccine, and GM-CSF After 11 patients have been assigned to each group, the study arm with the greatest number of vaccine-induced strong antibody responses will then continue with enrollment of 15 further patients. The primary objective is to determine the best strategy to induce strong (>15 fold) tumor-specific or tumor-associated antibody responses in patients with stage III A and B NSCLC. The goal is to select one regimen to advance to additional clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Stage IIIA or IIIB histologically proven non-small cell lung cancer
* Completion of definitive therapy
* Enrollment from 28 days to 12 weeks from completion of definitive therapy
* Toxicities from definitive therapy resolved to less than grade 1
* ECOG performance status 0-1
* Negative pregnancy test in women of childbearing potential
* Agree to avoid pregnancy or fathering a child while on study treatment
* Ability to give informed consent and comply with protocol
* Anticipated survival minimum of 6 months
* Prior therapy with investigational agents must be completed at least 3 weeks prior to study enrollment
* Normal organ and marrow function as defined by specific lab tests
* Archived tumor tissue available

Exclusion Criteria:

* Active autoimmune disease except for vitilogo or hypothyroidism
* Active other malignancy
* Known HIV+ and/or Hepatitis B or C positive
* Medical or psychiatric conditions that would preclude safe participation
* Ongoing chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-07; Primary Completion 2016-11 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Identify the regimen that produces the strongest antibody response | 95 days
  The best regimen will be defined as the one that generates the greatest increase in the number of strong antibody responses as defined by a greater than 15-fold increase in antibody, as measured using the Immune Response Biomarker Profiling Array (Invitrogen) on the day 95 serum sample.

SECONDARY OUTCOMES:
Safety | 43 weeks
  To evaluate the overall safety of allogeneic NSCLC DRibble vaccine alone or in combination with either imiquimod or GM-CSF, as adjuvant treatment for definitively-treated patients with Stage IIIA or B NSCLC. During the treatment period, patients will be seen in clinic 13 times over a 22-week period; performance status and side-effects will be evaluated at each visit.
Progression free survival | 2 years
  Evaluate progression-free survival. Tumor measurements by CT scan will be obtained at week 16 and subsequently at the discretion of the treating investigator. After the treatment period, patients will be seen every 3 months for 2 years, or until progressive disease.
Immune response and progression-free survival correlation. | 2 years
  Evaluate whether any immune response data correlate with progression-free survival. Immune response data will be collected 12 times over the first 43 weeks and then every 3 months until two years or progressive disease. This data will be correlated with progression-free survival.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Fox, PhD, Study Director — UbiVac
Locations (2):
- United States (2):
  - LSU Stanley S. Scott Cancer Center, New Orleans, Louisiana
  - Providence Cancer Center, Portland, Oregon